CLINICAL TRIAL: NCT00375739
Title: A Multi-center, Randomized, Double-blind, Double-dummy, Vehicle-controlled Sequential Cohort Study to Determine the Safety PEP005 0.025% and 0.05% Topical Gel in Patients With Actinic Keratoses.
Brief Title: Study to Determine the Safety of PEP005 0.025% and 0.05% Topical Gel in Patients With Actinic Keratoses
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peplin (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: PEP005-006
Record Dates: First submitted 2006-09-11; First posted 2006-09-13 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Actinic Keratosis
Keywords: Actinic Keratosis; Topical; Solar Keratosis; Sun Spots; Dermatology
MeSH Terms: conditions — Keratosis, Actinic; Melanosis | interventions — 3-ingenyl angelate

INTERVENTIONS:
Drug: PEP005

SUMMARY:
The purpose of this study is to determine whether topical application of PEP005 is safe for the treatment of actinic keratoses.

DETAILED DESCRIPTION:
Actinic keratoses (AK) is a common skin condition characterized by rough, scaly patches or sores on the top layer of the skin which if left untreated can progress to skin cancer. Current treatments can cause scarring and hypopigmentation, be inconvenient, or require long treatment duration. Non-invasive alternative therapy for treatment of AK lesions is thus being researched.

ELIGIBILITY:
Inclusion

1. Male patients at least 18 years of age.
2. Post-menopausal female patients i.e., no menses for at least 12 consecutive months, or without a uterus.
3. 4 to 8 clinically typical, visible and discrete AK lesions within a contiguous 25 cm2 treatment area on the arm, shoulder, chest, back or scalp.
4. Screening laboratory values within the reference ranges as defined by the central laboratory or "out of range" test results that are clinically acceptable to the Investigator.
5. Ability to follow study instructions and likely to complete all study requirements.
6. Written informed consent has been obtained.
7. Written Authorization for Use and Release of Health and Research Study Information has been obtained.
8. Agreement from the patient to allow photographs of the selected AK treatment area to be taken and used as part of the study data package.

Exclusion

1. Females of child bearing potential (a female is considered of childbearing potential unless she is postmenopausal, i.e., no menses for at least 12 consecutive months, or is without a uterus).
2. Location of the selected AK treatment area:

   1. anywhere on the face
   2. within 5 cm of an incompletely healed wound
   3. on the breast area of women
   4. on the dorsum of the hand
3. AK lesions that have atypical clinical appearance e.g. hypertrophic, hyperkeratotic, recalcitrant disease (had cryosurgery on 2 previous occasions), cutaneous horns within the selected AK treatment area.
4. Presence of suspected basal cell carcinoma (BCC) or squamous cell carcinoma (SCC) within the selected AK treatment area or within 10 cm of the selected AK treatment area.
5. Presence of known or suspected metastatic disease.
6. History or evidence of skin conditions other than AK that would interfere with evaluation of the study drug (e.g. eczema, unstable psoriasis, xeroderma pigmentosa).
7. Known sensitivity to any of the ingredients in the study drug.
8. A cosmetic or therapeutic procedure (e.g. use of liquid nitrogen, surgical excision, curettage, dermabrasion, medium or greater depth chemical peel, laser resurfacing):

   * within 2 cm of the selected AK treatment area during the 4 weeks prior to screening visit
9. Treatment with 5-fluorouracil, imiquimod, diclofenac, masoprocol or photodynamic therapy:

   * within 2 cm of the selected AK treatment area during the 24 months prior to screening visit or
   * anywhere during the 4 weeks prior to screening visit
10. Treatment with other immunomodulators (e.g. vinblastine, podophyllin, colhamin, camptothecin), cytotoxic drugs (e.g. cyclophosphamide, azathiopine, chlorambucil, nitrogen mustard, methotrexate), or interferon/ interferon inducers:

    * within 4 weeks prior to screening visit
11. Use of acid-containing therapeutic products (e.g. salicylic acids or fruit acids, such as alpha and beta hydroxy acids and glycolic acids), topical retinoids or light chemical peels:

    * within 2 cm of the selected AK treatment area during the 4 weeks prior to screening visit
12. Treatment with psoralen plus UVA (PUVA) or use of UVB therapy:

    * anywhere during the 6 months prior to screening visit
13. Use of systemic retinoids (e.g. isotretinoin, acitretin, bexarotene):

    * within 6 months prior to screening visit
14. Anticipated excessive or prolonged exposure to ultraviolet light (e.g. sunlight, tanning beds).
15. Use of topical salves, artificial tanners or topical steroids:

    * On the selected AK treatment area during the 4 weeks prior to screening visit
16. Anticipated need for hospitalization (in-patient) or surgery (except that specified in exclusion criteria 8) during the study.
17. Concurrent disease that suppresses the immune system (e.g. HIV, hepatitis).
18. Uncontrolled systemic disease (e.g. uncontrolled hypertension [a systolic blood pressure of 180 mmHg or greater and/or a diastolic blood pressure of 110 mmHg or greater], poorly controlled diabetes [fasting blood sugar of 350 mg/dl or greater]).
19. Use of systemic medications that suppress the immune system (e.g. cyclosporine, prednisone, methotrexate, alefacept, infliximab):

    * within 4 weeks prior to screening visit
20. Current evidence of chronic alcohol or drug abuse.
21. Current enrollment in an investigational drug or device study or participation in such a study within 30 days of entry into this study or entry into another investigational drug or device study while enrolled in this study.
22. A condition or situation which in the Investigator's opinion may put the patient at significant risk, may confound the study results, or may interfere significantly with the patient's participation in the study [e.g. patients who required hospitalization in the 2 months prior to screening for an acute or chronic condition].
23. Selected AK treatment area within 5 cm of an AK lesion previously treated with PEP005, for those patients who have participated in earlier PEP005 topical gel trials. Patients enrolled in Treatment Phase 1 can not be re-enrolled into Treatment Phase 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2006-09; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Safety

SECONDARY OUTCOMES:
Resolution of AK

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Anderson, Dr, Principal Investigator; Peter Welburn, PhD, Study Chair — Sponsor GmbH
Locations (24):
- United States (24):
  - Medical Affiliated Research Center, Inc., Huntsville, Alabama
  - Radiant Research, Tucson, Arizona
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Advanced Dermatology and Cosmetic Surgery, Clermont, Florida
  - Dermatology Associates and Research, Coral Gales, Florida
  - North Florida Dermatology Associates P.A., Jacksonville, Florida
  - Park Avenue Dermatology, PA, Orange Park, Florida
  - Dermatology Associates of Tallahassee, Tallahassee, Florida
  - Palm Beach Aesthetics, West Palm Beach, Florida
  - Medaphase, Inc, Newnan, Georgia
  - Gwinnett Clinical Research Centre, Inc, Snellville, Georgia
  - Henry Ford Health Center- Farmington Road, West Bloomfield, Michigan
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - St. Luke's/Roosevelt Hospital Center Dermatology, New York, New York
  - Mount Sinai Hospital School of Medicine, New York, New York
  - University Dermatology Consultants, Inc., Dermatology Clinical Research Center, Cincinnati, Ohio
  - Radiant Research, Columbus, Ohio
  - Oregon Medical Research, Centre9495 Southwest Locust St., Suite G Portland, Oregon
  - Radiant Research, Anderson, South Carolina
  - Radiant Research, Greer, South Carolina
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - Dermatology Associates of Tyler, Tyler, Texas
  - Dermatology Research Centre, Salt Lake City, Utah
  - Skokane Dermatology Clinic, PLLP., Spokane, Washington